CLINICAL TRIAL: NCT04414969
Title: Anti-PD-1 Antibody, Peg-Asparaginase, Chidamide Combined With Radiotherapy for the First-line Treatment of Patients With Stage I/II Extranodal Natural Killer/T Cell Lymphoma, Nasal Type (ENKTL): An Open-label, Multicenter, Phase II Trial
Brief Title: Anti-PD-1 Antibody Combined With Peg-Asparaginase and Chidamide for the Early Stage of NK/T Cell Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hunan Cancer Hospital (Other)
Responsible Party: Principal Investigator, Ya-Jun Li, Sub-Investigator, Hunan Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HNCH-NKT-2020
Record Dates: First submitted 2020-05-31; First posted 2020-06-04 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Immune Checkpoint Inhibitor; Chemotherapy Effect; Epigenetic Disorder; NK/T-cell Lymphoma of Nasal Cavity

STUDY DESIGN:
Intervention Model Description: An Open-label, multicenter, single group, phase II trial,
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anti-PD-1 antibody+Peg-Asparaginase+Chidamide (Experimental): Anti-PD-1 antibody 200mg ivdrip d1; PEG-ASP 2500U/m2 im d1; Chidamide, 30mg, PO, on d1，d5，d8，d12，d15，d19; repeat every 3 weeks.
  Interventions: Drug: Anti-PD-1 antibody+Peg-Asparaginase+Chidamide

INTERVENTIONS:
Drug: Anti-PD-1 antibody+Peg-Asparaginase+Chidamide — Anti-PD-1 antibody 200mg ivdrip d1, PEG-ASP 2500U/m2 im d1, Chidamide, 30mg, po, on d1，d5，d8，d12，d15，d19. The regimen was repeated every 3 weeks for 4 cycles followed by involved-field radiotherapy after got CR and PR (patients with efficacy of SD and PD withdrew from the study). Intensity-modulated radiation treatment was done by linear accelerator at 2.0 grays (Gy) per daily fraction with 5-6 weeks. The involved- field radiation (IFRT) dose was 54-56 Gy. During the radiotherapy, the anti-PD-1 antibody is administrated (200mg ivdrip, every 3 weeks) for 2 cycles. After the completion of radiotherapy, the subsequent 2 cycles of anti-PD-1 antibody + Peg-Asparaginase + Chidamide are administrated. After the end of all the above induction treatments , anti-PD-1 antibody (200mg ivdrip, every 3 weeks for up to 9 cycles) is given as maintenance therapy for 6 months (the total cycles of anti-PD-1 antibody is 17）.
  Other Names: Anti-PD-1 antibody；Peg-Asparaginase；Chidamide

SUMMARY:
This prospective pilot study to evaluate the efficacy and safety of the anti-PD-1 antibody combine with Peg-asparaginase and Chidamide regimen for stage IE and IIE ENKTL.

DETAILED DESCRIPTION:
Extranodal natural killer/T-cell lymphoma (ENKTL) is an aggressive subtype of non-Hodgkin's lymphoma and shows extremely poor survival. Several retrospective studies and randomized prospective phase 2 studies have shown that Peg-aspargase based chemotherapy regimens achieved a promising efficacy in the first line treatment of ENKTL. However, about one third of patients will relapse or become refractory after Peg-aspargase-based chemotherapy followed by radiotherapy, and some patients cannot tolerate the toxicities caused by chemotherapy. Anti-PD-1/PD-L1 antibodies and Chidamide are active drugs for the treatment of relapsed/refractory ENKTL. However, there is no prospective study to evaluate the efficacy and safety of anti-PD-1 antibody combine with Peg-asparaginase and Chidamide in the newly diagnosed early stage ENKTL. This prospective pilot study to evaluate the efficacy and safety of the anti-PD-1 antibody combine with Peg-asparaginase and Chidamide regimen for stage IE and IIE ENKTL.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically confirmed, previously untreated ENKTL with stage I/II (for stage I, the patients should have one or more of the following risk factors: ①Extensive local invasion and or bone destruction: invasion of the inner orbital wall or bottom wall, orbital apex, orbital contents, maxillary sinus, sphenoid sinus, frontal sinus or ethmoid sinus invasion, hard palate, ethmoid plate, nasopharynx, slope bone is invaded. ②Skin invasion: nose and or cheek skin invasion; ③Waldeyer's ring invasion; ④LDH>upper limit of normal; ⑤EBV-DNA > upper limit of normal; ⑥B symptoms);
2. Age range from 18 to 75 years;
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2;
4. At least one evaluable or measurable lesion complying with Lugano 2014 Standard (evaluable lesion: the examination show increased uptake of lymph nodes or extranodal areas (higher than that of the liver) by 18F-Fluorodeoxyglucose/Positron Emission Tomography (18FDG/PET) and the PET and/or Computed Tomography (CT) features coincide with lymphoma characteristics; measurable lesion: nodal lesions were longer than 15 mm or extranodal lesions were longer than 10 mm, and accompanied by increased 18FDG uptake). Increased liver or spleen diffuse 18FDG uptake without measurable lesions should be excluded.
5. Adequate haematologic function (haemoglobin ≥90 g/l, absolute neutrophil count ≥ 1500/ml, platelets ≥ 80×10e9/l),
6. Adequate hepatic function (total serum bilirubin ≤ 1.5 times the upper limit of normal, alanine aminotransferase and aspartate aminotransferase ≤ 2.5 times the upper limit of normal),
7. Hepatitis B virus carriers should have HBV-DNA <10e4 copies and should use antiviral drugs.
8. Adequate renal function (serum creatinine ≤ 1.5 mg/dl, creatinine clearance ≥ 50 ml/min);
9. Normal coagulation function and electrocardiogram results.
10. No previous anti-cancer treatment including chemotherapy, radiotherapy, immunotherapy, biological therapy, glucocorticoids therapy for lymphoma.
11. Willingness to provide written informed consent.

Exclusion Criteria:

1. History of other malignancy within the past 5 years (except for basal cell carcinoma of the skin and carcinoma in situ of the cervix)
2. With clinically diagnosed hemophagocytic syndrome (HPS); or aggressive NK cell leukemia; or central nervous system invasion;
3. Previous treatments with immune checkpoint inhibitor, including nivolumab, pembrolizumab, atezolizumab, durvalumab, avelumab, ipilimumab, sintilimab, etc.
4. Previous treatments with HDAC inhibitor, including Chidamide, romidepsin, panobinostat, belinostat, etc.
5. Patients allergic of any of drug in this regimen;
6. Pregnant or lactating women
7. Participated in other clinical trials within the 4 weeks prior to enrollment;
8. History of severe hemorrhage, or any bleeding events with a severe grade of 3 or more in CTCAE 5.0 within 4 weeks prior to enrollment
9. Blood pressure unable to be controlled ideally with single antihypertensive drug therapy (Systolic blood pressure > 140 mmHg, Diastolic Blood Pressure > 90 mmHg); Clinically significant cardiovascular disease (e.g. activity) including history of CVA (within 6 months), myocardial infarction (within 6 months), unstable angina, New York Heart Association (NYHA) Grade II or greater congestive heart failure; serious cardiac arrhythmia beyond drug control or potentially affecting experimental therapy.
10. The subject is being treated with immunosuppressive agents, glucocorticoids （systemic or absorbable local using）for immunosuppression purposes (dose> 10 mg / day prednisone or other therapeutic glucocorticoids) within two weeks before enrollment the study.
11. Abnormal coagulation or bleeding tendency (It must be satisfied that INR is under normal range without anticoagulant within 14 days prior to signing informed consent); patients treated with anticoagulants or vitamin K antagonists such as warfarin, heparin or their analogues; on the premise that the international standardized ratio of prothrombin time (INR) is less than 1.5, small doses of warfarin (1 mg po, qd) or aspirin (no more than 100 mg qd) are allowed for preventive purposes.
12. Arterial or venous thromboembolic events occurred within 6 months, such as cerebrovascular accident (including transient ischemic attack), deep vein thrombosis (venous thrombosis caused by intravenous catheterization due to precancerous chemotherapy is excluded if it has been cured judged by the researchers) and pulmonary embolism.
13. Suffered major surgery within 42 days prior to enrollment;
14. Have an active autoimmune disease that requires systemic treatment within the past two years.
15. Severe or uncontrolled infections, except fever associated with lymphoma B symptoms.
16. History of psychotropic drug abuse and unable to get rid of or with mental disorders;
17. History of immunodeficiency, including HIV positive testing, or other acquired, congenital immunodeficiency disorders, or organ transplantation history;
18. Patients with concomitant diseases which could seriously endanger their own safety or could affect completion of the study according to investigators' judgment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2020-06-26 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 12 weeks after the initiation of the treatment
  complete remission rate + partial remission rate
Complete remission rate | 12 weeks after the initiation of the treatment
  complete remission rate

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | Up to three years after the start of the study
  Time from the date of enrollment to date of disease progression, or death of any cause, or date of lost follow-up, whichever comes first, otherwise subject data were censored at time last known disease free.
Overall Survival (OS) | Up to three years after the start of the study
  Time from the date of enrollment to date of death from any cause, or date of lost follow-up, whichever comes first, and otherwise censored at time last known alive.
Safety issue | Up to one year after the end of the study
  All the adverse events of the patients related will be assessed and graded by NCI CTCAE v 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Hui Zhou, M.D., Principal Investigator — Department of Lymphoma and Hematology, Hunan Cancer Hospital
Locations (1):
- Hunan Cancer Hospital, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No